CLINICAL TRIAL: NCT07025863
Title: Construction and Application of an Intervention Program for Alarm Fatigue Among NICU Nurses Based on the ABC-X Theoretical Model
Brief Title: Intervention Program for Alarm Fatigue in NICU Nurses Based on ABC-X Model
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Guizhou Medical University (Other)
Collaborators: The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024282
Record Dates: First submitted 2025-06-09; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-03

CONDITIONS: Alert Fatigue, Health Personnel
Keywords: Neonatal Intensive Care Unit; Alarm Fatigue; ABC-X Model
MeSH Terms: conditions — Alert Fatigue, Health Personnel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): This study employed a self-control before-and-after experimental design. The aim is to initially apply the NICU nurse alarm fatigue intervention program based on the ABC-X theoretical model. By evaluating the implementation effect of the intervention and the satisfaction of the nurses, the effectiveness of the program will be verified and the program will be improved.
  Interventions: Behavioral: Alarm Fatigue Intervention Program

INTERVENTIONS:
Behavioral: Alarm Fatigue Intervention Program — Train nurses in terms of alarm fatigue stressors, coping resources, and cognition. The training content for stress management includes forming a multidisciplinary team, selecting appropriate equipment, replacing accessories and dressings in a timely manner, and comforting the children promptly. The training content for dealing with resources includes standardizing alarm response procedures, increasing manpower allocation, enhancing knowledge, skills, and psychological adjustment, etc. The training content of cognition includes fostering a positive attitude and strengthening responsibility, etc.

SUMMARY:
Monitors in newborn intensive care (NICU) help keep babies safe, but the constant beeping can overwhelm nurses. This 'alarm fatigue' makes it harder for nurses to identify real emergencies, stresses them out, and can impact patient care, including infant care. While we know this problem exists, there aren't many proven solutions. This study aims to develop and evaluate a new support program for nurses in the NICU who experience alarm fatigue. We first talked to NICU nurses to understand their challenges and needs. Then, using a stress management model (called the ABC-X model), we designed a program specifically to help them cope. Experts helped refine the program. Finally, we'll introduce this program to NICU nurses and see how well it works. The goal is to reduce nurses' alarm fatigue, improve their well-being, and ultimately enhance the safety and quality of care for newborns.

DETAILED DESCRIPTION:
Title: Construction and Application of an Intervention Program for Alarm Fatigue Among NICU Nurses Based on the ABC-X Theoretical Model

Background: Alarm fatigue in Neonatal Intensive Care Units (NICUs) is a critical patient safety and healthcare workers' well-being issue. The proliferation of monitoring technologies generates excessive, often clinically insignificant alarms, leading to desensitization, delayed responses, missed critical events, increased stress, burnout, and reduced quality of care among nurses. Current research primarily focuses on describing and quantifying alarm fatigue, with a significant gap in theory-driven intervention programs designed to mitigate its effects specifically for NICU nurses.

Objective: To develop, refine, and preliminarily apply a structured intervention program aimed at reducing alarm fatigue among NICU nurses, utilizing the ABC-X family stress model as a theoretical framework.

Methods: This study employs a multi-phase, sequential design:

Problem Exploration & Needs Assessment (Phase 1):

Literature Analysis: A systematic review of existing evidence on alarm fatigue causes, consequences, and interventions in NICUs.

Semi-Structured Interviews: In-depth interviews will be conducted with a purposive sample of NICU nurses to explore their lived experiences, perceptions, specific stressors, coping mechanisms, and perceived needs related to alarm management and fatigue.

Program Construction (Phase 2):

Theoretical Framework: The ABC-X model will guide program development. This model conceptualizes stress (X) as the outcome of a stressor event (A-e.g., alarm burden) interacting with the family's/resources (B-e.g., coping skills, unit support) and the perception (C-e.g., threat appraisal) of that event. The intervention will target modifiable A (stressors), B (resources), and C (perceptions/appraisals) factors.

Draft Intervention: Based on Phase 1 findings and ABC-X theory, an initial multi-component intervention program will be formulated. Potential components could include strengthening alarm management and improving physiology; cognitive-behavioral strategies for stress appraisal and coping; skills training (e.g., alarm customization, prioritization); environmental/organizational modifications; and peer support structures.

Delphi Expert Consultation: The draft program will be refined through iterative rounds of review using the Delphi method. A panel of experts (e.g., experienced NICU nurses, nurse managers, clinical nurse specialists, psychologists, neonatologists, and biomedical engineers) will independently rate and provide feedback on the program's components, feasibility, relevance, and potential effectiveness until consensus is achieved.

Program Application & Preliminary Evaluation (Phase 3):

The finalized intervention program will be implemented with a group of NICU nurses.

The application process will involve delivering the program components (e.g., workshops, training sessions, support groups, environmental adjustments) according to the developed protocol.

The feasibility of implementation and preliminary effects on nurses' levels of alarm fatigue (using validated scales), nurse clinical alert knowledge, attitude, and behavior, and satisfaction will be assessed.

Significance: By rigorously constructing an intervention rooted in the ABC-X stress model and refining it through expert consensus, the resulting program has the potential to provide a practical and scientific framework for healthcare institutions to mitigate alarm fatigue, thereby enhancing nurse well-being and patient safety in the vulnerable NICU population.

ELIGIBILITY:
Inclusion Criteria:

* Be informed and agree to participate in this study
* Have worked continuously in the NICU for at least 1 year
* Be a registered nurse with a practicing qualification certificate

Exclusion Criteria:

* Rotate and train nurses
* Those who are not on duty during the research period
* Those who did not directly participate in clinical work
* Those who withdrew from the research voluntarily during training
* Those whose attendance rate was less than 90% due to personal reasons

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
the level of alarm fatigue | Baseline and 1 week after intervention
  The Nurses' Alarm Fatigue Questionnaire (NAFQ) was developed by Iranian scholars Torabizadeh et al. in 2017 and is currently one of the most widely used self-assessment tools for quantifying the degree of alarm fatigue among ICU nurses. Chinese scholars Liu Jie et al. translated this questionnaire in 2021. It consists of 13 items, each using a 5-point Likert scale, with scores ranging from 0 to 4 representing "always, often, occasionally, very rarely, never," respectively. Items 1 and 9 are positively scored, while the remaining items are negatively scored. The total score ranges from 0 to 52 points, with higher scores indicating more severe alarm fatigue among ICU nurses. The Chinese version of the scale has a Cronbach's α coefficient of 0.771, a test-retest reliability of 0.966, and a content validity of 0.920, demonstrating good reliability and validity.

SECONDARY OUTCOMES:
The NICU Nurse Alarm Fatigue Intervention Program Satisfaction | 1 week after intervention
  The NICU Nurse Alarm Fatigue Intervention Program Satisfaction Survey Form will be used. This study designed its intervention satisfaction survey form, which includes intervention content, intervention methods, intervention class hours, learning difficulty, intervention quality, guidance significance for clinical practice, and overall evaluation. The evaluation results include very dissatisfied, dissatisfied, average, satisfied, and very satisfied. Satisfaction = (number of satisfied respondents + number of very satisfied respondents) / total number of respondents × 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Li, Principal Investigator — Guizhou Medical University
Locations (1):
- Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying study results will be shared. This includes:
  Quantitative survey responses (score on the Nurses' Alarm Fatigue Questionnaire) Aggregated qualitative themes from interviews (not raw transcripts) Demographic variables (age, gender, position, education, work experience) What data will NOT be shared? Audio recordings/raw interview transcripts (to protect participant confidentiality) Hospital identifiers or unit-specific performance metrics Personnel records of participating nurses
Supporting Information: Study Protocol, SAP
Time Frame: Following final publication of primary results (anticipated within 12 months of study completion).
Access Criteria: Researchers providing:
  * Approved ethics protocol
  * Signed data use agreement upon direct request to the principal investigator.